CLINICAL TRIAL: NCT00507923
Title: Effects of Tibetan Yoga on Fatigue and Sleep in Cancer
Brief Title: Tibetan Yoga in Improving Fatigue and Sleep in Participants With Stage I-III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-0035; NCI-2018-01753 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2005-0035 (Other: M D Anderson Cancer Center); R01CA105023 (NIH)
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Breast Cancer
Keywords: Breast Cancer; Tibetan Yoga; Stretching; Yoga; Fatigue; Sleep; Questionnaire; Survey
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Practice Guidelines as Topic; Standard of Care; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Tibetan yoga) (Experimental): Participants participate in Tibetan yoga sessions consisting of deep breathing or stretching exercises over 90 minutes for 4 sessions either once weekly or every 3 weeks. Participants also wear actigraph activity monitor and complete a sleep diary for 7 days. Participants receive instructional yoga audiotape and printed instructions to use at home upon completion of sessions.
  Interventions: Device: Actigraph; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Sleep Diary; Procedure: Yoga
- Group II (stretching) (Active Comparator): Participants participate in stretching exercise sessions over 90 minutes for 4 sessions either once weekly or every 3 weeks. Participants also wear actigraph activity monitor and complete a sleep diary for 7 days. Participants receive instructional yoga audiotape and printed instructions to use at home upon completion of sessions. Participants have the option to attend Tibetan yoga sessions upon completion of 12-month follow-up.
  Interventions: Device: Actigraph; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Sleep Diary; Other: Stretching
- Group III (usual care) (Active Comparator): Participants receive usual care and wear actigraph activity monitor and complete a sleep diary for 7 days. Participants have the option to attend Tibetan yoga sessions upon completion of 12-month follow-up.
  Interventions: Device: Actigraph; Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Sleep Diary

INTERVENTIONS:
Device: Actigraph — Wear actigraph
  Other Names: Actigram
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group III (usual care)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Sleep Diary — Complete sleep diary
  Other Names: Sleep Journal; Sleep Log
Other: Stretching — Participate in stretching sessions
  Arms: Group II (stretching)
Procedure: Yoga — Participate in Tibetan yoga
  Other Names: Yoga Therapy
  Arms: Group I (Tibetan yoga)

SUMMARY:
The goal of this behavioral research study is to learn if participating in a Tibetan yoga program helps to improve quality of life for women during treatment for or recovery from breast cancer. Researchers are also interested in whether the yoga program helps to improve sleep, lung function, and physical therapy, based on outcomes.

DETAILED DESCRIPTION:
You will come to M. D. Anderson for an initial meeting. You will complete several questionnaires asking about mood, quality of life, and other things like sleep, fatigue, anxiety, and coping skills. You will also have an electrocardiogram (ECG - a test to measure the electrical activity of your heart). Both the questionnaires and the ECG test should take about 60 minutes, total, to complete.

You will also wear an actigraph (a watch-like instrument that records arm movements) for 7 days. The actigraph records information about your physical activity, rest, and sleep. You will be asked to complete daily sleep diary forms that ask about some behaviors, your sleep, and sleep quality for the 7 days. At the end of the 7 days, you will return the actigraph and sleep diaries to the research staff, or a member of the research staff can go to your home to pick them up.

If you are assigned to the yoga group, you will take part in 4 weekly sessions of Tibetan yoga. If you are not able to attend 4 weekly sessions, you can attend 1 session every 3 weeks, for a total of 4 sessions over 12 weeks, of Tibetan yoga. You will be asked to complete a brief form at the start of each session that will take 1-2 minutes to complete. During the yoga sessions, you will be asked to do deep breathing exercises and perform different stretching and movement exercises. You will be able to move through the exercises at your own pace. Sessions occurring weekly will last 90 minutes. Sessions occurring once every 3 weeks will last 90 minutes. All sessions will be provided free of charge. One or more of these yoga sessions may be videotaped by the study staff for quality assurance purposes. Only the study staff will be able to view this videotape.

If you are assigned to the stretching group, you will take part in 4 weekly sessions in which you will be asked to do simple stretching exercises. If you are not able to attend 4 weekly sessions, you can attend 1 session every 3 weeks, for a total of 4 sessions over 12 weeks. Sessions occurring weekly will last 90 minutes. Sessions occurring once every 3 weeks will last 90 minutes. All sessions will be provided free of charge. None of the movements are difficult. You will be able to follow this program at your own pace.

If you are assigned to the yoga or stretching group, you will take part in 3 "booster" sessions consisting of a review and practice of the entire program. If you are in the 4 weekly sessions, your booster sessions will take place 1 and 2 months after your last yoga or stretch class and again around the time of your 6-month assessment. If you are in the classes that meet every 3 weeks over a 12-week period, your booster sessions will take place 3 and 6 weeks after your last yoga or stretch class and again around the time of your 6-month assessment.

If a need for counseling/therapy arises, your primary care physician will be notified and can refer you to the Section of Psychiatry, Department of Neuro-Oncology.

One week, 3 months, 6 months, and 12 months after the end of the yoga or stretching sessions (or similar time for the usual care group), you will be asked to return to the clinic. You will fill out a packet of questionnaires and complete an ECG evaluation again. The questionnaires and tests should take about 60 minutes to complete. You will also be asked to wear the actigraph and complete daily sleep diary forms for another 7 days. At the end of the 7 days, you will return the actigraph and sleep diaries to the research staff, or a member of the research staff can go to your home to pick them up. This will be your last participation in the study.

After the study is over, if you took part in the stretching or were in the usual care group, you will be given the option to take the yoga classes.

ELIGIBILITY:
Inclusion Criteria:

1. Women with stage I-III breast cancer who are undergoing neoadjuvant or adjuvant chemotherapy weekly for 12 weeks followed by four cycles of an anthracycline-based treatment every 21 days or six to eight cycles of chemotherapy every 21 days or are within 24 months post-treatment (surgery and/or chemotherapy and/or radiotherapy - patients can still be taking hormonal treatment).
2. 18 years of age or older.
3. Able to read, write and speak English
4. Able to come to UTMDACC for intervention and assessment sessions.

Exclusion Criteria:

1. Metastatic disease of the bone.
2. Documented diagnosis of a formal thought disorder (e.g., schizophrenia).
3. Engaged in psychiatric or psychological counseling or support groups.
4. Reports the need for psychological services.
5. Score of 23 or below on the Mini-Mental State Examination.
6. Presence of lymphedema at the start of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2006-11-07 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
The correlation on the effects of Tibetan yoga on fatigue | Up to 12 months
  Participants will be monitored on the extent to which the Tibetan Yoga program decreases fatigue and sleep disturbances. Fatigue will be assessed using the Brief Fatigue Inventory (BFI). The BFI is a 9-item questionnaire designed to be used in the clinical setting to rapidly assess fatigue severity. The items are ranked from 0 to 10, and patients rate their fatigue at its "worst" and "usual" and as it is "now," with 0 = "no fatigue" and 10 = "fatigue as bad as you can imagine." Patients also rate how much their fatigue has interfered with their life. This single-dimension instrument was tested in a sample of patients with cancer, and provided an internally stable measure of fatigue severity.
The correlation on the effects of Tibetan yoga on sleep disturbances | Up to 12 months
  The Fatigue will be assessed using the Brief Fatigue Inventory (BFI), items are ranked from 1-10 and patients will rate their fatigue at its "worst" and "usual" and as it is "now" with 0= no fatigue and 10= "fatigue as bad as you can imagine". The Sleep disturbance will be assessed using the Pittsburgh Sleep Quality Index (PSQI), this 18 item questionnaire and it rates the sleep quality from 0=good and 3=very poor. The less the total score the less of a sleep disturbance problem.
Identifying the process of the underlying efficacy of Tibetan yoga intervention. | Up to 12 months
  Writing will be conducted at the 3 month post intervention assessment. Participants will only conduct the writing one time as an outcome measure, which should not have an appreciable affect on the outcomes. Samples will be analyzed using Linguistic Inquiry Word Count (LIWC) software was developed to examine the linguistic content of writing samples. We used this program in our previous pilot study examining the emotional-expression writing intervention. The software counts the number of times specific words are used in the writing samples. The software recognizes more than 2,290 words and classifies them into 74 different grammatical, cognitive, and emotional categories. It can calculate the average percentage of words used in the different categories and determine changes in the percentages over writing samples. Writings will also be assessed in an exploratory fashion using qualitative analyses, including the use of ethnographic methods.
The Effects of Tibetan Yoga Program with the aspects of adjustment. | Up to 12 months
  We will assess cytotoxicity to K562 target cells; stimulated and circulating release of IL-12, IFN, IL-4, IL-6, IL-8, and IL-10 (using polyclonal stimulators); flow cytometric analysis of intracellular cytokines (to identify the subset of cells producing the particular cytokine); and lymphocyte phenotype (CD3, CD56, CD16, CD4, and CD8) [279, 280]. PBMCs will be cryopreserved for future analyses if the initial assays are encouraging. Other assays may be conducted in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org